CLINICAL TRIAL: NCT02207400
Title: A Six Month Clinical Study Based in the US to Evaluate the Efficacy and Tolerability of Sodium Bicarbonate Toothpaste and Its Effect on Opportunistic or Resistant Organisms
Brief Title: To Evaluate Efficacy and Tolerability of Sodium Bicarbonate Toothpaste and Its Effect on Opportunistic or Resistant Organisms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202193; RH02434 (Other: GSK)
Record Dates: First submitted 2014-07-21; First posted 2014-08-04 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Sodium Bicarbonate; Sodium Fluoride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Dentifrice (Experimental): Participants were advised to brush their teeth with experimental dentifrice containing sodium bicarbonate plus 1150 parts per million (ppm) fluoride as sodium fluoride
  Interventions: Drug: Sodium bicarbonate and sodium fluoride
- Reference Dentifrice (Active Comparator): Participants were advised to brush their teeth with reference dentifrice containing 1100ppm fluoride as sodium fluoride
  Interventions: Drug: Sodium fluoride

INTERVENTIONS:
Drug: Sodium bicarbonate and sodium fluoride — Experimental toothpaste containing sodium bicarbonate experimental dentifrice plus 1150 parts per million (ppm) fluoride as sodium fluoride
  Arms: Experimental Dentifrice
Drug: Sodium fluoride — Comparator toothpaste containing 1100 ppm fluoride as sodium fluoride
  Arms: Reference Dentifrice

SUMMARY:
This study will compare the Gingival Bleeding and Gingival Inflammation following twice daily use of a sodium bicarbonate experimental dentifrice compared to a 0% sodium bicarbonate toothpaste after 24 weeks of use. The study will be conducted at Salus Research, Inc. Participants will be recruited from their database and by use of an external recruitment agency

DETAILED DESCRIPTION:
This study will be a single-centre, examiner blind, two treatment, parallel group, stratified (by baseline number of bleeding sites smoking status and bacterial sampling) randomized clinical study. At the screening visit, following provision of written informed consent, eligible participants will be provided with a standard toothpaste and toothbrush for brushing once in at the clinic and for approximately one week use at home until the baseline visit. Participants will be asked to abstain from brushing over a 12 hour period prior to the Baseline visit. At the baseline visit an oral soft tissue (OST) assessment, Modified Gingival Index (MGI) and Bleeding Index (BI), and then dental plaque assessment will be performed. Participants will be stratified according to their baseline number of bleeding sites, smoking status and whether selected for bacterial sampling. Participants will be then randomized into one of two treatment groups. After using, their assigned treatment twice daily at home for 6 weeks (visit 3), 12 weeks (visit 4) and 24 weeks (visit 5), participants will return to the site with overnight plaque at approximately the same time of day as the Baseline visit if possible. Participants will undergo a full OST examination and the recording of any Adverse Events (AEs). Participants will then undergo MGI, BI followed by dental plaque assessment. Microbiological samples will be collected on a subset of 50 participants (Determined by first 50 participants randomized).

ELIGIBILITY:
Inclusion Criteria:

* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral/dental examination.
* A minimum of 20 permanent gradable teeth
* Moderate gingivitis present at the screening visit in the opinion of the investigator
* A total of 20 bleeding sites or greater at baseline visit
* Positive response to bleeding on brushing present at the screening visit

Exclusion Criteria:

* Pregnant or breast feeding women
* Tobacco chewers
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any other medical condition (e.g. Diabetes Mellitus) that would make the participant unlikely to fully complete the study or any that increases the risk to the participant or undermines the data validity.
* Recent history (within the last year) of alcohol or other substance abuse
* Participants requiring prophylactic antibiotic treatment prior to dental therapy
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Have current active caries or any medical conditions which may directly influence gingival bleeding
* Use of concomitant or any systemic medication that, in the opinion of the investigator, might interfere with the outcome of the study or have an effect on gingival conditions within 14 days of gingival examinations
* Excessive calculus present that interferes with the probing examination for Gingival Bleeding Index
* Participation in another clinical study or receipt of an investigational drug or oral care product within 30 days of the screening visit
* An employee of the sponsor or the study site or members or their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

REFERENCES:
- [Derived] Jose A, Pratten J, Bosma ML, Milleman KR, Milleman JL, Wang N. Six-Month Evaluation of a Sodium Bicarbonate-Containing Toothpaste for Reduction of Established Gingivitis: A Randomized USA-Based Clinical Trial. J Clin Dent. 2018 Mar;29(1):33-39. PMID 29758155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited at a clinical site in the USA.
Groups:
- Sodium Bicarbonate and Sodium Fluoride Dentifrice: Experimental toothpaste containing sodium bicarbonate experimental dentifrice plus 1150 parts per million (ppm) fluoride as sodium fluoride
- Sodium Fluoride Dentifrice: Toothpaste containing 1100 ppm fluoride as sodium fluoride
Period: Overall Study
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Started | 123 | 123
Completed | 107 | 109
Not Completed | 16 | 14
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 6 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Positive Urine Pregnancy Test | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice | Total
Number analyzed (Participants) | 123 | 123 | 246
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.39 (14.284) | 37.77 (12.615) | 38.58 (13.473)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 152
  Male | 49 | 45 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Gingival Bleeding Sites at 24 Weeks
Description: The Bleeding Index was performed by a single examiner using a color coded periodontal probe. The probe was engaged approximately 1 millimetre (mm) into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed
Time Frame: 24 weeks
Population: ITT population defined as those participants who had received study treatment and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Number of bleeding sites
Groups:
- Sodium Bicarbonate and Sodium Fluoride Dentifrice: Experimental dentifrice containing sodium bicarbonate plus 1150 parts per million (ppm) fluoride as sodium fluoride
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
Number of bleeding sites | 13.24 (7.663) | 24.90 (9.044)
Statistical Analysis 1: Comparison: Sodium Bicarbonate and Sodium Fluoride Dentifrice vs Sodium Fluoride Dentifrice; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted Mean Difference = -11.612, 95% CI 2-sided [-13.191 to -10.033] — Difference is Sodium Bicarbonate and Sodium Fluoride Dentifrice minus Sodium Fluoride Dentifrice such that a negative difference favors the first named treatment

2. Primary Outcome: Modified Gingival Index (MGI) at 24 Weeks
Description: MGI was assessed on facial and lingual surfaces at two sites on each tooth (papillae and margin). The scoring of the MGI was performed under dental office conditions using a standard dental light for illuminating the oral cavity. Compressed air, water and mouth mirrors were available to each examiner. This procedure was performed by a single examiner. The MGI scoring system is as follows: 0 = absence of inflammation; 1 = mild inflammation; slight change in color, little change in color; little change in texture of any portion of the marginal or papillary gingival unit; 2 = mild inflammation; criteria as above but involving the entire marginal or papillar gingival units; 3= moderate inflammation; glazing, redness, edema, and/ or hypertrophy of the marginal or papillary gingival unit; 4 = severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Sodium Bicarbonate and Sodium Fluoride Dentifrice: Experimental dentifrice containing sodium bicarbonate plus 1150 ppm fluoride as sodium fluoride
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
Units on a scale | 1.26 (0.505) | 1.93 (0.408)
Statistical Analysis 1: Comparison: Sodium Bicarbonate and Sodium Fluoride Dentifrice vs Sodium Fluoride Dentifrice; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.652, 95% CI 2-sided [-0.738 to -0.566] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Gingival Bleeding Sites at 6 and 12 Weeks
Description: BI was performed by a single examiner using a color coded periodontal probe. The probe was engaged approximately 1mm into the gingival crevice. A moderate pressure was used whilst sweeping from interproximal to interproximal along the sulcular epithelium. The BI scoring system used is as follows: 0= No bleeding after 30 seconds; 1= Bleeding upon probing after 30 seconds; 2= Immediate bleeding observed
Time Frame: Baseline, 6 and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of bleeding sites
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
Number of bleeding sites
  Number of Bleeding Sites at Baseline | 29.76 (8.238) | 29.05 (8.390)
  Number of Bleeding Sites at 6 weeks | 12.26 (9.339) | 23.23 (10.993)
  Number of Bleeding Sites at 12 weeks | 15.73 (7.632) | 23.86 (9.265)

4. Secondary Outcome: Modified Gingival Index (MGI)) at 6 and 12 Weeks.
Description: as for outcome 2
Time Frame: 6 and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
Units on a scale
  MGI at 6 weeks | 1.50 (0.567) | 1.96 (0.427)
  MGI at 12 weeks | 1.50 (0.536) | 1.94 (0.464)

5. Secondary Outcome: Bleeding Index (BI) at 6, 12 and 24 Weeks
Description: as for outcome 3
Time Frame: 6, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
Units on a Scale
  BI Score Score at 6 weeks | 0.15 (0.133) | 0.30 (0.172)
  BI Score Score at 12 weeks | 0.19 (0.112) | 0.28 (0.135)
  BI Score Score at 24 weeks | 0.17 (0.116) | 0.31 (0.159)

6. Secondary Outcome: Plaque Control (Overall and Interproximal Dental Plaque Scores) at 6, 12 and 24 Weeks.
Description: The dental examiner had used the Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth. Interproximal Dental Plaque Scores were analyzed in the same way as for Overall scores but just based on mesiofacial, facial, distofacial, mesiolingual, lingual and distolingual surfaces. Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5: 0= No plaque; 1= Slight flecks of plaque at the cervical margin of the tooth; 2= A thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3= A band of plaque wider than 1 mm but covering less than 1/3 of the crown of the tooth; 4= Plaque covering at least 1/3 but less than 2/3 of the crown of the tooth; 5= Plaque covering 2/3 or more of the crown of the tooth.
Time Frame: 6, 12 and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Sodium Bicarbonate and Sodium Fluoride Dentifrice: Experimental toothpaste containing sodium bicarbonate experimental dentifrice plus 1150 ppm fluoride as sodium fluoride
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 112
Units on a scale
  Overall Plaque Score at 6 weeks | 2.56 (0.536) | 3.01 (0.411)
  Overall Plaque Score at 12 weeks | 2.54 (0.495) | 2.90 (0.374)
  Overall Plaque Score at 24 weeks | 2.47 (0.437) | 2.92 (0.399)
  Interproximal Plaque Score at 6 weeks | 2.78 (0.492) | 3.19 (0.351)
  Interproximal Plaque Score at 12 weeks | 2.76 (0.437) | 3.10 (0.311)
  Interproximal Plaque Score at 24 weeks | 2.71 (0.390) | 3.11 (0.336)

7. Secondary Outcome: Bacterial Count at Baseline, After 6, 12, 24 and 32 Weeks
Description: Microbiological samples were collected at baseline, 6 weeks, 12 weeks, 24 weeks and 32 weeks. Plaque was harvested from contra-lateral 1st molar teeth, where no restorations are present, using a sterile paper point. The paper point was immersed into 4 ml of Calgon Ringer's solution in a sterile bijou and kept on ice until they can be taken to the laboratory for processing (within 24 hours).
Time Frame: Baseline, 6, 12, 24 and 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: colony forming units per sample
Groups:
- Sodium Bicarbonate and Sodium Fluoride Dentifrice: Experimental toothpaste containing sodium bicarbonate experimental dentifrice plus 1150 ppm)fluoride as sodium fluoride
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Number analyzed (Participants) | 118 | 117
colony forming units per sample
  Staph Count at Baseline (n=24, 26) | 0.2 (0.82) | 0.2 (0.86)
  Steph Count at 6 weeks (n=24, 26) | 0.1 (0.34) | 0 (0.20)
  Steph Count at 12 weeks (n=24, 26) | 1.8 (7.10) | 3.2 (15.47)
  Steph Count at 24 weeks (n=23, 25) | 0.6 (1.59) | 0.2 (0.37)
  Steph Count at 32 weeks (n=21, 21) | 0.2 (0.51) | 0.1 (0.36)
  Yeast Count at Baseline (n=24, 26) | 203.4 (842.28) | 647.8 (2958.78)
  Yeast Count at 6 weeks (n=23, 26) | 287.3 (1014.31) | 784.3 (1796.75)
  Yeast Count at 12 weeks (n=24, 25) | 668.9 (812.81) | 411.3 (906.19)
  Yeast Count at 24 weeks (n=17, 22) | 1479.6 (1165.48) | 1522.3 (1008.13)
  Yeast Count at 32 weeks (n= 14, 14) | 2743.5 (2505.75) | 1206.4 (1008.34)
  Coliform count at Baseline (n= 24, 26) | 3.9 (8.82) | 3.8 (8.27)
  Coliform count at 6 weeks (n= 24, 26) | 2.6 (6.72) | 5.7 (20.05)
  Coliform count at 12 weeks (n= 24, 26) | 10.9 (14.65) | 26.9 (78.47)
  Coliform count at 24 weeks (n=23, 25) | 8.1 (16.86) | 12.6 (19.24)
  Coliform count at 32 weeks (n=21, 21) | 10.9 (16.17) | 17.8 (29.84)
  E. Coli count at Baseline (n=24, 26) | 0 (0) | 0 (0.20)
  E. Coli count at 6 weeks (n=24, 26) | 0.1 (0.28) | 0 (0.20)
  E. Coli count at 12 weeks (n=24, 26) | 0.1 (0.28) | 0 (0)
  E. Coli count at 24 weeks (n=23, 25) | 0.3 (1.25) | 0.2 (0.55)
  E. Coli count at 32 weeks (n=21, 21) | 0.6 (1.29) | 0 (0.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study from the start of the washout period, until five days following last treatment.
Arm/Group | Sodium Bicarbonate and Sodium Fluoride Dentifrice | Sodium Fluoride Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/123
Other Adverse Events (participants affected / at risk) | 17/123 | 14/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate and Sodium Fluoride Dentifrice (N=123) | Sodium Fluoride Dentifrice (N=123)
Cellulitis Orbital (Infections and infestations) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
MOUTH INJURY (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (2)
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 (1) | 1 (1)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GINGIVAL ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TONGUE ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 1 (1) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.